CLINICAL TRIAL: NCT02802761
Title: Nutritional Assessment Tool in Childhood Chronic Liver Disease
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-CLD-Nutrition-02
Record Dates: First submitted 2016-03-21; First posted 2016-06-16 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-05

CONDITIONS: Chronic Liver Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Study Cohort:

All Children (Age: 3 months- 18 years, corrected age upto 2 years for preterm children) with Chronic Liver Disease attending Pediatric Hepatology Out Patient Department/In Patient Department

ELIGIBILITY:
Inclusion Criteria:

1. Children from age of 3 months- 18 years (corrected age upto 2 years for preterm children)
2. Chronic liver disease.

Exclusion Criteria:

1. Any metabolic or endocrinal diseases independently affecting nutritional status
2. Refusal to give written informed consent to participate in the study

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All Children (Age: 3 months to 18 years, corrected age upto 2 years for preterm children) with CLD attending Pediatric Hepatology OPD/IPD.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Reliability of SGNA versus nutritional status as assessed by standard anthropometric measures in children with chronic liver disease. | 2 years
  Nutritional status (well nourished, moderate or severe malnutrition) of a child with chronic liver disease as assessed by standard anthropometric measures (weight, height, mid arm circumference, Body mass index, triceps and subscapular skin fold thickness) will be compared to the results of nutritional assessment score as obtained by applying Subjective Global Nutritional Assessment (SGNA) proforma.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Seema Alam, MD, Study Director — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided